CLINICAL TRIAL: NCT00652483
Title: Safety and Efficacy Study of Brimonidine in Patients With Glaucoma or Ocular Hypertension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Therapeutic Area Head, Allergan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 190342-021
Record Dates: First submitted 2008-04-01; First posted 2008-04-03 (Estimated); Last update posted 2008-04-03 (Estimated); Status verified 2008-04

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Brimonidine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Brimonidine ophthalmic solution 0.1%
  Interventions: Drug: Brimonidine ophthalmic solution 0.1%
- 2 (Active Comparator): Brimonidine ophthalmic solution 0.2%
  Interventions: Drug: Brimonidine ophthalmic solution 0.2%

INTERVENTIONS:
Drug: Brimonidine ophthalmic solution 0.1% — 1 drop instilled in each eye 3 times daily (08:00, 14:00, 20:00)
  Arms: 1
Drug: Brimonidine ophthalmic solution 0.2% — 1 drop instilled in each eye 3 times daily (08:00, 14:00, 20:00)
  Other Names: ALPHAGAN®
  Arms: 2

SUMMARY:
This study evaluates the safety and efficacy of brimonidine 0.1% ophthalmic solution compared with brimonidine 0.2% ophthalmic solution in patients with glaucoma or ocular hypertension

ELIGIBILITY:
Inclusion Criteria:

* Ocular hypertension or glaucoma in both eyes

Exclusion Criteria:

* Uncontrolled systemic disease
* Known allergy or sensitivity to brimonidine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 433 (Actual)
Dates: Start 2003-05; Primary Completion 2003-12 (Actual); Study Completion 2004-09 (Actual)

PRIMARY OUTCOMES:
Intraocular pressure (IOP) | Week 2 - Month 3

SECONDARY OUTCOMES:
IOP | Month 6 - Month 12

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Allergan
Locations (1):
- Atlanta, Georgia, United States

REFERENCES:
- See also: Link to Clinical Trial Results — http://www.allerganclinicaltrials.com